CLINICAL TRIAL: NCT01495598
Title: A Phase I/II Study of the Safety, Pharmacokinetics and Efficacy of Pomalidomide (CC-4047) in the Treatment of Kaposi Sarcoma in Individuals With or Without HIV
Brief Title: Pomalidomide for Kaposi Sarcoma in People With or Without HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 120047; 12-C-0047
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Kaposi Sarcoma; Sarcoma, Kaposi
Keywords: Human Herpesvirus-8/HHV8; Immune Modulation; CC-4047; IMiD; Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Pomalidomide 5mg Daily (Experimental): Up to six subjects will initially be treated with for 21 days of a 28 day cycle
  Interventions: Drug: Pomalidomide
- Phase 2 Pomalidomide 5mg Daily (Experimental): 15 human immunodeficiency virus (HIV) positive and 10 HIV negative subjects evaluable for response will be treated with Pomalidomide 5mg daily for 21 days of a 28 day cycle
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — 5 mg by mouth (p.o.) for 21 of 28 days
  Other Names: POMALYST®

SUMMARY:
Background:

- Pomalidomide is a drug that can treat cancer through several mechanisms. It is taken by mouth (orally). Pomalidomide can help treat cancer by blocking certain factors that promote tumor growth or by stimulating the immune system to attack tumor cells. It also prevents the growth of new blood vessels that help cancer grow. Researchers want to see if pomalidomide can treat Kaposi sarcoma, a rare and potentially fatal skin cancer. Because Kaposi sarcoma may be associated with human immunodeficiency virus (HIV) infection, researchers want to test the drug in people with and without HIV infection.

Objectives:

- To see if pomalidomide is a safe and effective treatment for Kaposi sarcoma in people with or without HIV.

Eligibility:

* Individuals at least 18 years of age who have Kaposi sarcoma.
* Participants may or may not have HIV infection.

Design:

* Potential participants will be screened with a medical history and physical exam. Blood and saliva samples will be taken and a chest X-ray will be performed. A skin biopsy of a Kaposi sarcoma lesion may be performed if one has not already been done. Other imaging studies may be performed if needed.
* Participants will take pomalidomide capsules every day for 3 weeks, followed by a 1-week break. These 28 days are one cycle of treatment.
* Participants will have up six cycles of treatment, unless the lesions completely resolve sooner. If there are signs of improvement after six cycles but the lesions are not completely gone, up to another six cycles of treatment may be given.
* Treatment will be monitored with frequent blood tests and other studies including photograph and other imaging of skin lesions.
* Participants will have regular follow-up visits for 5 years after stopping treatment....

DETAILED DESCRIPTION:
Background:

Kaposi Sarcoma (KS) is an incurable, multicentric angioproliferative tumor that most frequently involves the skin. It is seen most frequently in people with human immunodeficiency virus (HIV) or other forms of immune compromise. Current therapies are limited by toxicities, including cumulative cardiotoxicity, while effective oral agents, agents deliverable in resource-limited settings, and agents deliverable long-term for relapsing disease are all lacking.

Objective:

The primary objective of this study is to:

Assess the safety, tolerability and pharmacokinetics of pomalidomide in subjects with Kaposi sarcoma, whether HIV associated or not.

Eligibility:

* Age greater than or equal to 18 years
* Measurable, pathologically confirmed KS
* Any HIV status; HIV-associated KS subjects must be receiving and able to comply with highly active antiretroviral therapy (HAART) and have achieved an HIV viral load <10,000 copies/mL
* Hematologic and biochemical parameters within prespecified limits at baseline
* Willing to use effective birth control, as defined in the full protocol
* For subjects enrolled in the anti-tumor activity assessment phase, if KS is HIV-associated it must be increasing despite HAART and HIV suppression for greater than or equal to 2 months, or stable despite HAART for greater than or equal to 3 months
* No symptomatic pulmonary or visceral KS
* No specific KS therapy within 4 weeks (6 weeks if that therapy was bevacizumab)
* Neither pregnant nor breast feeding

Design:

This is an open label single agent phase I/II study of pomalidomide in patients with KS. In the phase I portion, up to six subjects will initially be treated with pomalidomide 5mg daily for 21 days of a 28 day cycle. Subject to toxicity evaluation, this dosage may be deescalated to 3mg daily for 21 days of a 28 day cycle in a second cohort of up to six subjects. If either dose proves tolerable, the study will proceed to the phase II portion, and additional subjects to a goal of 15 HIV positive and 10 HIV negative subjects evaluable for response will be added at the highest tolerable dose to gain preliminary information on activity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 Years.
* Any human immunodeficiency virus (HIV) status.
* Kaposi sarcoma pathologically confirmed by Department of Pathology, Clinical Center, National Institutes of Health.
* At least five measurable Kaposi sarcoma (KS) lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion.
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2
* Life expectancy greater than or equal to 6 months
* For patients with HIV-associated KS:

  * Must be receiving, and adherent to, a highly active antiretroviral therapy (HAART) regimen consistent with current clinical guidelines.
  * Must have been receiving HAART for at least one month.
  * Must have achieved an HIV viral load (VL) <10,000 copies/mL.
* The following hematological parameters:

  * Hemoglobin greater than or equal to 10 g/dL
  * Platelets greater than or equal to 75,000 cells/mm(3)
  * Absolute neutrophil count (ANC) greater than or equal to 1000 cells/mm(3)
* The following biochemical parameters:

  * Estimated or measured creatinine clearance greater than or equal to 45mL/minute
  * Serum alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal
  * Serum aspartate aminotransferase (AST) less than or equal to 2.5 times upper limit of normal
  * Bilirubin less than or equal to 1.5 times upper limit of normal unless the patient is receiving protease inhibitor therapy (e.g., indinavir, ritonavir, nelfinavir, or atazanavir) known to be associated with increased bilirubin, in which case total bilirubin less than or equal to 7.5 mg/dL with direct fraction less than or equal to 0.7 mg/dL.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 14 days prior to and again within 24 hours before starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, and also
* All study participants must agree to be registered into the mandatory POMALYST Risk Evaluation and Mitigation Strategy (REMS) program and be willing and able to comply with the requirements of the POMALYST REMS program.
* Females of reproductive potential must be willing to adhere to the scheduled pregnancy testing as required in the POMALYST REMS program.
* Able to take aspirin 81mg daily or if intolerant of aspirin, able to take a substitute thromboprophylaxis such as low molecular weight heparin at a thromboprophylactic dose (such as enoxaparin 0.5mg/kg once daily).
* Willing and able to give informed consent.
* For subjects with HIV-associated entered after a tolerable dose has been determined, KS lesions must be either:

  * Increasing despite HAART and HIV suppression below the limit of detection (48 copies/mL) in the two months prior to screening or
  * Stable despite HAART for at least three months. Stable disease must be symptomatic (examples of symptomatic disease include disease associated with pain, edema, psychological distress and/or social withdrawal). This is to gain preliminary information about pomalidomide activity without confounding due to HAART initiation.

EXCLUSION CRITERIA:

* Symptomatic pulmonary KS.
* Symptomatic visceral KS (except for non-ulcerating disease restricted to the oral cavity).
* Specific KS therapy, including cytotoxic chemotherapy but not including HAART, within the past 4 weeks (6 weeks if the therapy was bevacizumab).
* Use of other anticancer treatments or agents within the past 4 weeks (6 weeks if the therapy was a monoclonal antibody).
* History of malignant tumors other than KS, unless:

  * In complete remission for greater than or equal to 1 year from the time response was first documented or
  * Completely resected basal cell carcinoma or
  * In situ squamous cell carcinoma of the cervix or anus.
* History of infection meeting any of the following criteria:

  * Any infection that would be scored as grade 4 by Common Terminology Criteria for Adverse Events (CTCAE) that occurred within six weeks of study screening.
  * Any infection that would be scored as grade 3 by CTCAE that occurred within two weeks of study screening.
  * History of fungal and mycobacterial infections, unless at least six weeks has passed since the completion of induction antimicrobial therapy. Patients may be receiving consolidation therapy for infections of these types.
* Any abnormality that would be scored as a greater than or equal to grade 3 toxicity by CTCAE, except:

  * Obesity is not considered an abnormality for the purposes of eligibility assessment unless in the opinion of the Principal Investigator or Lead Associate Investigator its clinical consequences in a particular subject places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study.
  * Lymphopenia
  * Asymptomatic hyperuricemia, hypophosphatemia, or creatine kinase (CK) Elevations
  * Direct manifestations of KS
  * Direct manifestations of HIV infection, except for neurologic or cardiac manifestations
  * Direct manifestations of HIV therapy, except for neurologic or cardiac manifestations.
* History of venous or arterial thromboembolism, unless:

  * Line-related thrombosis without embolus occurring greater than or equal to 1 year prior to screening.

Complications resulting from atherosclerotic coronary artery disease, peripheral vascular disease, or cerebrovascular disease (including infarction) are not considered exclusion criteria unless in the opinion of the Principal Investigator or Lead Associate Investigator their clinical consequences in a particular subject places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study

* Known drug-related, inherited, or acquired procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome.
* Pregnancy.
* Breast feeding (if lactating, must agree not to breast feed while taking pomalidomide).
* Prior therapy with pomalidomide.
* Known hypersensitivity to thalidomide, lenalidomide or pomalidomide. including prior development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide or pomalidomide.
* Any condition, including the presence of laboratory abnormalities, which in the opinion of the Principal Investigator or Lead Associate Investigator places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. All collected IPD will be available after primary analysis have been published.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Krown SE. AIDS-associated Kaposi's sarcoma: pathogenesis, clinical course and treatment. AIDS. 1988 Apr;2(2):71-80. No abstract available. PMID 3132950
- [Background] Chang Y, Cesarman E, Pessin MS, Lee F, Culpepper J, Knowles DM, Moore PS. Identification of herpesvirus-like DNA sequences in AIDS-associated Kaposi's sarcoma. Science. 1994 Dec 16;266(5192):1865-9. doi: 10.1126/science.7997879.
- [Background] Uldrick TS, Whitby D. Update on KSHV epidemiology, Kaposi Sarcoma pathogenesis, and treatment of Kaposi Sarcoma. Cancer Lett. 2011 Jun 28;305(2):150-62. doi: 10.1016/j.canlet.2011.02.006. Epub 2011 Mar 4. PMID 21377267
- [Background] Feinberg J, Saag M, Squires K, Currier J, Ryan R, Coate B, Mrus J. Health-related quality of life in the gender, race, and clinical experience trial. AIDS Res Treat. 2011;2011:349165. doi: 10.1155/2011/349165. Epub 2011 Aug 28. PMID 21904672
- [Background] Cianfrocca M, Lee S, Von Roenn J, Tulpule A, Dezube BJ, Aboulafia DM, Ambinder RF, Lee JY, Krown SE, Sparano JA. Randomized trial of paclitaxel versus pegylated liposomal doxorubicin for advanced human immunodeficiency virus-associated Kaposi sarcoma: evidence of symptom palliation from chemotherapy. Cancer. 2010 Aug 15;116(16):3969-77. doi: 10.1002/cncr.25362. PMID 20564162
- [Background] Uldrick TS, Wang V, O'Mahony D, Aleman K, Wyvill KM, Marshall V, Steinberg SM, Pittaluga S, Maric I, Whitby D, Tosato G, Little RF, Yarchoan R. An interleukin-6-related systemic inflammatory syndrome in patients co-infected with Kaposi sarcoma-associated herpesvirus and HIV but without Multicentric Castleman disease. Clin Infect Dis. 2010 Aug 1;51(3):350-8. doi: 10.1086/654798. PMID 20583924
- [Result] Polizzotto MN, Uldrick TS, Wyvill KM, Aleman K, Peer CJ, Bevans M, Sereti I, Maldarelli F, Whitby D, Marshall V, Goncalves PH, Khetani V, Figg WD, Steinberg SM, Zeldis JB, Yarchoan R. Pomalidomide for Symptomatic Kaposi's Sarcoma in People With and Without HIV Infection: A Phase I/II Study. J Clin Oncol. 2016 Dec;34(34):4125-4131. doi: 10.1200/JCO.2016.69.3812. Epub 2016 Oct 31. PMID 27863194
- [Result] Ramaswami R, Polizzotto MN, Lurain K, Wyvill KM, Widell A, George J, Goncalves P, Steinberg SM, Whitby D, Uldrick TS, Yarchoan R. Safety, Activity, and Long-term Outcomes of Pomalidomide in the Treatment of Kaposi Sarcoma among Individuals with or without HIV Infection. Clin Cancer Res. 2022 Mar 1;28(5):840-850. doi: 10.1158/1078-0432.CCR-21-3364. PMID 34862247
- [Derived] Lurain K, Polizzotto MN, Krug LT, Shoemaker G, Singh A, Jensen SMR, Wyvill KM, Ramaswami R, Uldrick TS, Yarchoan R, Sereti I. Immunophenotypic analysis in participants with Kaposi sarcoma following pomalidomide administration. AIDS. 2023 Sep 1;37(11):1693-1703. doi: 10.1097/QAD.0000000000003627. Epub 2023 Jun 19. PMID 37352498
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0047.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Pomalidomide 5mg Daily: All participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
Period: Overall Study
Arm/Group | Pomalidomide 5mg Daily
Started | 28
Completed | 14
Not Completed | 14
Not completed — Death during follow up period | 2
Not completed — Death on study | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.5 [44.9 to 61.3]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender male | 27
  Transgender male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28
Prior Kaposi Sarcoma (KS) Therapy [Count of Participants; unit: Participants]
  Prior systemic therapy | 22
  Liposomal doxorubicin | 14
  Paclitaxel | 8
  Radiotherapy | 9
  Immunomodulatory therapy | 3
  Interferon alpha | 5
  Local therapy | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grades 1-4 Adverse Events That Are Possibly, Probably, and/or Definitely Attributed to Pomalidomide
Description: Adverse events (AE's) that are possibly, probably, and/or definitely attributed to pomalidomide were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: During each cycle and 4 weeks after completing therapy, with any continuing AE's observed until resolution, approximately 124 months and 1 day.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1: Grade 1 is mild.
- Grade 2: Grade 2 is moderate.
- Grade 3: Grade 3 is severe.
- Grade 4: Grade 4 is life-threatening.
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 28 | 28 | 28 | 28
Participants
  Low white cell count | 21 | 10 | 1 | 0
  Febrile neutropenia | 0 | 0 | 1 | 0
  Neutropenia | 24 | 26 | 14 | 3
  Lymphocytopenia | 13 | 2 | 0 | 0
  Anemia | 16 | 4 | 0 | 0
  Thrombocytopenia | 16 | 0 | 0 | 0
  Fatigue | 17 | 2 | 0 | 0
  Infection | 0 | 7 | 1 | 0
  Constipation | 18 | 3 | 0 | 0
  Nausea | 10 | 0 | 0 | 0
  Elevated alanine aminotransferase (ALT) | 7 | 0 | 0 | 0
  Impaired concentration | 3 | 1 | 0 | 0
  Depression | 1 | 1 | 0 | 0
  Hypothyroidism | 3 | 3 | 0 | 0
  Rash | 18 | 6 | 1 | 0
  Vasculitis | 0 | 0 | 1 | 0

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time from day 1 of pomalidomide therapy until progression requiring a change in therapy, estimated using the Kaplan-Meier method. Progression was assessed using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Group criteria. Progressive disease (PD) involved a 25% or greater increase in total lesions, nodular lesion, or area of the five indicator lesions.
Time Frame: time from day 1 of pomalidomide therapy until progression requiring a change in therapy, an average of 9.97 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants: All participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
- HIV Positive Participants: HIV positive participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
- HIV Negative Participants: HIV negative participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | All Participants | HIV Positive Participants | HIV Negative Participants
Number analyzed (Participants) | 28 | 18 | 10
months | 10.2 [7.6 to 15.7] | 10.3 [4.8 to 21.9] | 9.4 [6.0 to 26.0]
Statistical Analysis 1: Comparison: HIV Positive Participants vs HIV Negative Participants; Test type: Other — Other = Kaplan Meier; p = 0.43, Log Rank

3. Primary Outcome: Maximal Plasma Concentration (Cmax) of Pomalidomide
Description: Plasma concentrations of pomalidomide were assayed using high-performance liquid chromatography with fluorescence detection with a lower limit of quantitation of 1 ng/mL and were recorded as observed values. A non-compartmental analysis was used to calculate plasma pharmacokinetic parameters (Pharsight, Mountain View, California).
Time Frame: At pre-dose, 1, 2, 3, 4, 6, and 8 hours after dose on Cycle 1 Day 1, and pre-dose, 1, 2, 3, 4, 6, 8, and 24 hours after dose on Cycle 1 Day 15.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- All Participants - Pomalidomide 5mg Daily: All participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
ng/mL
  Cycle 1 Day 1 | 53.1 (27.0)
  Cycle 1 Day 15 | 59.0 (29.6)

4. Primary Outcome: Time to Maximum Observed Serum Concentration of Pomalidomide (Cmax)
Description: Time to maximum observed serum concentration of Pomalidomide was reported.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
hours
  Cycle 1 Day 1 | 2.00 [1 to 8]
  Cycle 1 day 15 | 2.08 [1 to 8]

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) to the Last Timepoint (AUCLast)
Description: Area under the plasma concentration versus time curve (AUC) was calculated using the log-linear trapezoidal method. The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
hours*ng/mL
  Cycle 1 Day 1 | 466.5 (304)
  Cycle 1 Day 15 | 504.5 (325.9)

6. Primary Outcome: Area Under the Curve Extrapolated to Infinity (AUCinf)
Description: AUC is a measure of the serum concentration of Pomalidomide over time. It is used to characterize drug absorption. The AUC extrapolated to infinity was used, unless the percent extrapolated exceeded 25% in which case AUC to the last quantifiable time point (AUCLast) was used. The steady-state exposure on Day 15 of cycle 1 was calculated using AUCLast.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours*ng/ml
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
hours*ng/ml
  Cycle 1 Day 1 | 567.3 (423.2)
  Cycle 1 Day 15 | 805.3 (986.9)

7. Primary Outcome: Half-Life of Pomalidomide
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
hours
  Cycle 1 Day 1 | 6.85 (2.13)
  Cycle 1 Day 15 | 8.27 (6.61)

8. Secondary Outcome: Antitumor Effect of a Second Course of Pomalidomide
Description: Antitumor effect of pomalidomide was assessed at the established tolerated dose after a second course of pomalidomide. Kaposi sarcoma responses were assessed using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Group criteria. Complete Response (CR) required clinical resolution of all lesions and tumor-associated phenomenon with biopsy confirmation. Clinical Complete Response (cCR) is resolution of all lesions except for some residual pigmentation but who did not have a biopsy of a representative pigmented area. Partial Response (PR) required ≥ 50% decrease in the number of lesions and/or sum product of the diameters of marker lesions and/or nodularity of lesions, and no new lesions in previously uninvolved areas or criteria. Stable Disease (SD) was assessed for all participants who did not meet criteria doe CR, PR, or PD. And progressive disease (PD) involved a 25% or greater increase in total lesions, nodular lesion, or area of the five indicator lesions.
Time Frame: After completion of 2 cycles of therapy up to 48 weeks after the start of the second course of Pomalidomide
Population: 4/28 participants were eligible for a second course of pomalidomide at time of progression within 12 months of treatment cessation.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants - Pomalidomide 5mg Daily: All participants that received a second course of pomalidomide: 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 4
Participants
  Complete Response (CR) | 0
  Clinical Complete Response (CCR) | 0
  Partial Response (PR) | 2
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 0

9. Secondary Outcome: Antitumor Effect of a First Course of Pomalidomide
Description: Antitumor effect of pomalidomide was assessed at the established tolerated dose after a first course of pomalidomide. Kaposi sarcoma responses were assessed using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Group criteria. Complete Response (CR) required clinical resolution of all lesions and tumor-associated phenomenon with biopsy confirmation. Clinical Complete Response (cCR) is resolution of all lesions except for some residual pigmentation but who did not have a biopsy of a representative pigmented area. Partial Response (PR) required ≥ 50% decrease in the number of lesions and/or sum product of the diameters of marker lesions and/or nodularity of lesions, and no new lesions in previously uninvolved areas or criteria. Stable Disease (SD) was assessed for all participants who did not meet criteria doe CR, PR, or PD. And progressive disease (PD) involved a 25% or greater increase in total lesions, nodular lesion, or area of the five indicator lesions.
Time Frame: After completion of 2 cycles of therapy up to 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- All Participants - Pomalidomide 5mg Daily: All participants that received a first course of pomalidomide: 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
Participants
  Complete Response (CR) | 1
  Clinical Complete Response (CCR) | 3
  Partial Response (PR) | 16
  Stable Disease (SD) | 5
  Progressive Disease (PD) | 3

10. Secondary Outcome: Self-Reported Health-Related Quality of Life (HRQL) Instrument: Functional Assessment of Human Immunodeficiency Virus Infection (FAHI)
Description: Changes in quality of life in participants receiving pomalidomide. HRQL was analyzed using a mixed-model repeated-measures analysis for FAHI and the marginal homogeneity test for Kaposi sarcoma-specific questions such as physical well-being (PWB), emotional well-being (EWB), functional and global well-being (FGWB), social well-being (SWB), and cognitive functioning (CF). The range of possible scores for each subscale was as follows: PWB and EWB, 0 to 40; FGWB, 0 to 52; SWB, 0 to 32; CF, 0 to 12. The total FAHI score, with possible scores ranging from 0 to 176, was calculated as the sum of all five subscale values, with higher scores indicating better results. Questionnaires completed at early withdrawal visits were not included in the analyses.
Time Frame: Baseline, after 3 months of therapy, and after completion of therapy, up to 48 weeks
Population: Missing responses within questionnaire in category FAHI Total at baseline (n=21). And missing responses within questionnaire in category FAHI Total after completion of therapy (n=17).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; After 3 Months of Therapy; After Completion of Therapy: All participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | Baseline | After 3 Months of Therapy | After Completion of Therapy
Number analyzed (Participants) | 22 | 19 | 19
score on a scale
  FAHI Total: number analyzed (Participants) | 21 | 19 | 17
  FAHI Total | 123.0 (30.2) | 123.4 (28.4) | 118. (29.0)
  Physical well-being | 30.8 (8.7) | 31.3 (8.2) | 31.3 (9.1)
  Emotional well-being | 25.1 (7.6) | 27.7 (7.5) | 26.2 (7.7)
  Functional and global well-being | 34.4 (10.3) | 34.5 (10.1) | 32.9 (9.6)
  Social well-being | 22.1 (6.6) | 21.5 (7.8) | 20.9 (6.8)
  Cognitive functioning | 9.1 (2.7) | 8.5 (2.7) | 8.7 (2.3)

11. Secondary Outcome: Number of Participants Who Responded to Each Question on the Self-Reported Health-Related Quality of Life (HRQL): Kaposi Sarcoma (KS) - Specific Questions
Description: The number of participants responding to each question with the indicated responses is shown. Changes in quality of life in participants receiving pomalidomide. HRQL was analyzed using a mixed-model repeated-measures analysis and the marginal homogeneity test for Kaposi sarcoma-specific questions. Three supplemental questions addressing pain, swelling, and satisfaction with physical appearance was used to collect quality of life data.
Time Frame: Baseline, timepoint 1: after 3 months of therapy, and timepoint 2: 1 month after completion of therapy
Population: 22 participants were analyzed at baseline. 19/22 participants were evaluable and analyzed at timepoint 2 and timepoint 3 because the QOL data was not collected on the other three participants at those timepoints. Baseline n=22, timepoint 2 = 19, and timepoint 3 = 19. *Sum of two preceding columns. ϮSum of three preceding columns.
Measure: Count of Participants; unit: Participants
Groups:
- Not At All; A Little Bit; Little or None*; Somewhat; Quite a Bit; Very Much; Somewhat or MoreϮ: Response on the HRQL questionnaire.
Arm/Group | Not At All | A Little Bit | Little or None* | Somewhat | Quite a Bit | Very Much | Somewhat or MoreϮ
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22 | 22
Participants
  Pain has interfered with my normal work or activities at baseline | 10 | 3 | 13 | 2 | 5 | 2 | 9
  Pain has interfered with my normal work or activities - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Pain has interfered with my normal work or activities - timepoint 2: after 3 months of therapy | 7 | 5 | 12 | 5 | 1 | 1 | 7
  Pain has interfered with my normal work or activities timepoint 3:1month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Pain has interfered with my normal work or activities timepoint 3:1month after completion of therapy | 7 | 5 | 12 | 4 | 1 | 2 | 7
  I am satisfied with my physical appearance at baseline | 6 | 6 | 12 | 6 | 3 | 1 | 10
  I am satisfied with my physical appearance - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I am satisfied with my physical appearance - timepoint 2: after 3 months of therapy | 6 | 1 | 7 | 5 | 5 | 2 | 12
  I am satisfied with my physical appearance - timepoint 3: 1 month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I am satisfied with my physical appearance - timepoint 3: 1 month after completion of therapy | 3 | 2 | 5 | 5 | 8 | 1 | 14
  I have had swelling in my face, arms, or legs at baseline | 6 | 2 | 8 | 5 | 4 | 5 | 14
  I have had swelling in my face, arms, or legs - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I have had swelling in my face, arms, or legs - timepoint 2: after 3 months of therapy | 7 | 2 | 9 | 4 | 4 | 2 | 10
  I have had swelling in my face, arms, or legs - timepoint 3: 1 month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I have had swelling in my face, arms, or legs - timepoint 3: 1 month after completion of therapy | 6 | 3 | 9 | 4 | 5 | 1 | 10

12. Secondary Outcome: Change in Cytokines From Baseline to 4 Weeks, Baseline to 8 Weeks and End of Treatment
Description: Cytokines were evaluated using MSD 96-Well Multiarray Proinflammatory 7-plex assay (MesoScale Discovery).
Time Frame: Baseline to 4 weeks, baseline to 8 weeks and baseline to end of treatment
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Baseline to 4 Weeks: Baseline to 4 weeks for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
- Baseline to 8 Weeks: Baseline to 8 weeks for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
- Baseline to End of Treatment: Baseline to end of treatment for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days.
Arm/Group | Baseline to 4 Weeks | Baseline to 8 Weeks | Baseline to End of Treatment
Number analyzed (Participants) | 28 | 28 | 28
pg/mL
  Interferon gamma (ƴ) | -0.3 [-4.7 to 1.4] | -0.4 [-7.4 to 4.5] | -2.4 [-5.3 to 55.1]
  Interleukin 4 (IL4) | 0.07 [0.02 to 0.1] | 0.1 [0.04 to 0.2] | 0.06 [0.001 to 0.1]
  Interleukin 6 (IL6) | 0.4 [-0.04 to 1.8] | 0.3 [-0.3 to 1.1] | 0.6 [-0.3 to 5.8]
  Interleukin 8 (IL8) | 71.9 [5.3 to 163.1] | 64.8 [-0.2 to 233.1] | 47.5 [-9.1 to 121.1]
  Interleukin 10 (IL10) | 0.1 [-0.1 to 1.4] | -0.03 [-0.2 to 0.4] | -0.05 [-0.3 to 0.2]
  Interleukin 12 (IL12) | 0.02 [-0.08 to 0.09] | 0.00 [-0.07 to 0.09] | 0.03 [-0.07 to 0.14]
  Interleukin 13 (IL13) | 0.7 [0.03 to 1.9] | 0.9 [0.0 to 1.7] | 0.6 [-0.02 to 1.3]
  Tumor necrosis factor alpha (TNFα) | 0.3 [-0.09 to 0.8] | 0.5 [0.1 to 0.8] | 0.06 [-0.3 to 0.4]
  Interferon (IFN)-inducible protein 10 (IP-10) | 76.5 [-214.5 to 239.3] | 18.4 [-271.7 to 216.6] | -73.3 [-335.7 to 127.8]
Statistical Analysis 1: Comparison: Baseline to 4 Weeks; Test type: Other — <0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.19, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IFNƴ among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.72, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.03, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p < 0.0001, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL4 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p < 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 4]
Statistical Analysis 6: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p < 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 4]
Statistical Analysis 7: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.005, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL6 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 8: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.06, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 7]
Statistical Analysis 9: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.007, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 7]
Statistical Analysis 10: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.0003, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL8 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 11: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.0002, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 10]
Statistical Analysis 12: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.01, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 10]
Statistical Analysis 13: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.03, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 7]
Statistical Analysis 14: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.91, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL10 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 15: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.64, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 14]
Statistical Analysis 16: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.70, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL12 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 17: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.59, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 16]
Statistical Analysis 18: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.26, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 16]
Statistical Analysis 19: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.0008, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IL13 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 20: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p < 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 19]
Statistical Analysis 21: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.007, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 19]
Statistical Analysis 22: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.005, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of TNFα among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 23: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.007, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 22]
Statistical Analysis 24: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.007, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 22]
Statistical Analysis 25: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.42, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of IP-10 among all participants. Two tailed Wilcoxon signed rank test without adjustment for multiple comparisons
Statistical Analysis 26: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.85, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 25]
Statistical Analysis 27: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.16, Wilcoxon signed rank test — [p-value comment as in outcome 12, analysis 25]

13. Secondary Outcome: Change in Immune Cytokines Cluster of Differentiation 4 (CD4), Cluster of Differentiation 8 (CD8) and Cluster of Differentiation 19 (CD19) Among Participants With and/or Without Human Immunodeficiency Virus (HIV)
Description: Fluorescence activated cell sorting.
Time Frame: Baseline to 4 weeks, baseline to 8 weeks, and baseline to end of treatment
Population: HIV+ participants = 18.
Measure: Median (Inter-Quartile Range); unit: cells/µL
Groups:
- Baseline to 4 Weeks: Baseline to 4 weeks for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days. Includes 18 HIV+ participants.
- Baseline to 8 Weeks: Baseline to 8 weeks for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days. Includes 18 HIV+ participants.
- Baseline to End of Treatment: Baseline to end of treatment for participants treated with pomalidomide 5 mg by mouth (p.o.) for 21 of 28 days. Includes 18 HIV+ participants.
Arm/Group | Baseline to 4 Weeks | Baseline to 8 Weeks | Baseline to End of Treatment
Number analyzed (Participants) | 28 | 28 | 28
cells/µL
  CD4+/All participants | 66.5 [-77.5 to 221] | 37 [-57.0 to 176.0] | -54 [-178.5 to 91.5]
  CD4+ among HIV+ participants: number analyzed (Participants) | 18 | 18 | 18
  CD4+ among HIV+ participants | 72 [-29 to 257] | 37 [-15 to 291] | -14 [-79 to 132]
  CD8+/All participants | 104.5 [-76.5 to 257] | 115 [-19 to 288] | 73 [-38.5 to 194.5]
  CD8+ among HIV+ participants: number analyzed (Participants) | 18 | 18 | 18
  CD8+ among HIV+ participants | 198 [-20 to 414] | 129 [1 to 430] | 75 [-102 to 295]
  CD19+/All participants | -40 [-73 to -3.5] | -55 [-123 to 5] | -75 [-124.5 to -49.5]
Statistical Analysis 1: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.07, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD4+ cells/µL among all participants
Statistical Analysis 2: Comparison: Baseline to 8 Weeks; Test type: Non-Inferiority — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.13, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD4+cells/µL among all participants
Statistical Analysis 3: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.15, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD4+cells/µL among all participants
Statistical Analysis 4: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.03, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD4+cells/µL among HIV+ participants
Statistical Analysis 5: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.06, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD4+cells/µL among HIV+ participants
Statistical Analysis 6: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.79, Wilcoxon rank sum test — The reported p-value is representative of the changes in levels of CD4+cells/µL among HIV+ participants
Statistical Analysis 7: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.03, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among all participants
Statistical Analysis 8: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.008, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among all participants
Statistical Analysis 9: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.12, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among all participants
Statistical Analysis 10: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.02, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among HIV+ participants
Statistical Analysis 11: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.02, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among HIV+ participants
Statistical Analysis 12: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.36, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD8+ cells/µL among HIV+ participants
Statistical Analysis 13: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.002, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD19+ cells/µL among all participants
Statistical Analysis 14: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.0002, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD19+ cells/µL among all participants
Statistical Analysis 15: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p < 0.0001, Wilcoxon signed rank test — The reported p-value is representative of the changes in levels of CD19+ cells/µL among all participants

14. Secondary Outcome: Change Between Timepoints Baseline to 4 Weeks, Baseline to 8 Weeks, and Baseline to End of Treatment in Kaposi Sarcoma-Associated Herpesvirus (KSHV) Viral Load
Description: KSHV viral load in peripheral blood mononuclear cells was assessed by modifying a sandwich enzyme-linked immunosorbent assay (ELISA). Viral load testing may provide useful information on the occurrence of KSHV replication. Undetectable levels is good.
Time Frame: Baseline to 4 weeks, baseline to 8 weeks and baseline to end of treatment
Population: PBMC = peripheral mononuclear cells
Measure: Median (Inter-Quartile Range); unit: copies per million PBMC
Arm/Group | Baseline to 4 Weeks | Baseline to 8 Weeks | Baseline to End of Treatment
Number analyzed (Participants) | 28 | 28 | 28
copies per million PBMC | 0 [0 to 136] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.13, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.65, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.32, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.06, Wilcoxon signed rank test
Statistical Analysis 5: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.007, Wilcoxon signed rank test

15. Secondary Outcome: Human Immunodeficiency Virus (HIV) Viral Load
Description: HIV viral load in peripheral blood mononuclear cells was assessed by quantitative real-time polymerase chain reaction (PCR). The lower limit of detection for HIV viral load is <50 copies mL.
Time Frame: Baseline to 4 weeks, baseline to 8 weeks and baseline to end of treatment
Measure: Median (Inter-Quartile Range); unit: Copies/mL
Arm/Group | Baseline to 4 Weeks | Baseline to 8 Weeks | Baseline to End of Treatment
Number analyzed (Participants) | 28 | 28 | 28
Copies/mL | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Baseline to 4 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.56, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Baseline to 8 Weeks; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.65, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Baseline to End of Treatment; Test type: Other — P<0.005 was considered statistically significant while 0.005 <P<0.05 was considered evidence of a strong trend; p = 0.56, Wilcoxon signed rank test

16. Secondary Outcome: Percentage of Participants Who Responded to Each Question on the Self-Reported Health-Related Quality of Life (HRQL): Kaposi Sarcoma (KS) - Specific Questions
Description: The percentage of participants responding to each question with the indicated responses is shown. Changes in quality of life in participants receiving pomalidomide. HRQL was analyzed using a mixed-model repeated-measures analysis and the marginal homogeneity test for Kaposi sarcoma-specific questions. Three supplemental questions addressing pain, swelling, and satisfaction with physical appearance was used to collect quality of life data.
Time Frame: Baseline, timepoint 1: after 3 months of therapy, and timepoint 2: 1 month after completion of therapy
Population: 22 participants were analyzed at baseline. 19/22 participants were evaluable and analyzed at timepoint 2 and timepoint 3 because the QOL data was not collected on the other 3 participants at those timepoints. Baseline n=22, timepoint 2 = 19, and timepoint 3 = 19. *Sum of two preceding columns. ϮSum of three preceding columns.
Measure: Number; unit: percentage of participants
Arm/Group | Not At All | A Little Bit | Little or None* | Somewhat | Quite a Bit | Very Much | Somewhat or MoreϮ
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22 | 22
percentage of participants
  Pain has interfered with my normal work or activities at baseline | 45.5 | 13.6 | 59.1 | 9.1 | 22.7 | 9.1 | 40.9
  Pain has interfered with my normal work or activities - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Pain has interfered with my normal work or activities - timepoint 2: after 3 months of therapy | 36.8 | 26.3 | 63.2 | 26.3 | 5.3 | 5.3 | 36.8
  Pain has interfered with my normal work or activities timepoint 3:1month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Pain has interfered with my normal work or activities timepoint 3:1month after completion of therapy | 36.8 | 26.3 | 63.2 | 21.1 | 5.3 | 10.5 | 36.8
  I am satisfied with my physical appearance at baseline | 27.3 | 27.3 | 54.6 | 27.3 | 13.6 | 4.5 | 45.4
  I am satisfied with my physical appearance - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I am satisfied with my physical appearance - timepoint 2: after 3 months of therapy | 31.6 | 4.5 | 36.8 | 26.3 | 26.3 | 10.5 | 63.2
  I am satisfied with my physical appearance - timepoint 3: 1 month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I am satisfied with my physical appearance - timepoint 3: 1 month after completion of therapy | 15.8 | 10.5 | 26.3 | 26.3 | 42.1 | 5.3 | 73.7
  I have had swelling in my face, arms, or legs at baseline | 27.3 | 9.1 | 36 | 22.7 | 18.2 | 22.7 | 63.6
  I have had swelling in my face, arms, or legs - timepoint 2: after 3 months of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I have had swelling in my face, arms, or legs - timepoint 2: after 3 months of therapy | 36.8 | 10.5 | 47 | 21.1 | 21.1 | 10.5 | 52.6
  I have had swelling in my face, arms, or legs - timepoint 3: 1 month after completion of therapy: number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 19
  I have had swelling in my face, arms, or legs - timepoint 3: 1 month after completion of therapy | 31.6 | 15.8 | 47 | 21.1 | 26.3 | 5.3 | 52.6

17. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 124 months and 1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
Participants | 28

18. Other Pre Specified Outcome: Number of Dose-limiting Toxicities
Description: A dose limiting toxicity is any grade 4 toxicity not including lymphopenia, cluster of differentiation 4 (CD4) lymphopenia, neutropenia, anemia and bilirubin or creatine kinase (CK) elevation that is at least possibly due to pomalidomide and is not attributable to human immunodeficiency virus (HIV), its therapy or Kaposi Sarcoma (KS). Any grade 3 toxicity that is at least possibly due to pomalidomide and is not attributable to HIV, its therapy, or KS and restrictions such as grade 3 thrombocytopenia if grade 3 for 14 days or more, Grade 3 asymptomatic hyperuricemia or hypophosphatemia, or Grade 3 amylase elevations.
  Any arterial or deep venous thromboembolic event or a second superficial thromboembolic event that is at least possibly due to pomalidomide. Inability to deliver pomalidomide on at least 50% of scheduled days during the first two cycles of therapy as a result of toxicity that is probably or definitely attributable to pomalidomide.
Time Frame: First 8 weeks (2 cycles) of drug administration
Measure: Number; unit: toxicities
Arm/Group | All Participants - Pomalidomide 5mg Daily
Number analyzed (Participants) | 28
toxicities | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 124 months and 1 day.
Arm/Group | Pomalidomide 5mg Daily
All-Cause Mortality (participants affected / at risk) | 4/28
Serious Adverse Events (participants affected / at risk) | 12/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide 5mg Daily (N=28)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Death Not otherwise specified (NOS) (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Gastrointestinal disorders - Other, gastrointestinal (GI) bleed (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Anal squamous cell carcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Bladder tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Metastatic basaloid squamous cell carcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Scalp basal cell carcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Squamous cell carcinoma of skin right heel
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — basal cell carcinoma; Right Lower Back
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Vasculitis (Vascular disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide 5mg Daily (N=28)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 7 (9)
Alanine aminotransferase increased (Investigations) | 16 (47)
Alkaline phosphatase increased (Investigations) | 5 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Amylase (Investigations) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 22 (61)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 12 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 4 (6)
Blurred vision (Eye disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (13)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Cluster of differentiation (CD4) lymphocytes decreased (Investigations) | 12 (33)
Creatine phosphokinase (CPK) increased (Investigations) | 8 (28)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 5 (5)
Concentration impairment (Nervous system disorders) | 3 (7)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 21 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Creatinine increased (Investigations) | 10 (24)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 9 (21)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Edema face (General disorders) | 1 (3)
Edema limbs (General disorders) | 14 (26)
Edema trunk (General disorders) | 1 (1)
Enterocolitis (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - Other, Blepharitis (Eye disorders) | 1 (1)
Eye disorders - Other, excessive wetness (Eye disorders) | 1 (1)
Eye disorders - Other, left eye nodule (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 18 (54)
Fever (General disorders) | 5 (7)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, gastrointestinal (GI) distress (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, abdominal cramping (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Cramps in Lower extremities and arms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, Decreased appetite (General disorders) | 1 (1)
General disorders and administration site conditions - Other, Imbalance due to Hip Pain (General disorders) | 1 (2)
General disorders and administration site conditions - Other, Night Sweats (General disorders) | 1 (1)
Gum infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Hematuria (Renal and urinary disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (15)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 6 (7)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (44)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (10)
Hyponatremia (Metabolism and nutrition disorders) | 8 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 21 (83)
Hypothyroidism (Endocrine disorders) | 7 (9)
International normalized ratio (INR) increased (Investigations) | 1 (2)
Immune system disorders - Other, insect bite reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other, prominent insect bite (Immune system disorders) | 1 (1)
Infections and infestations - Other, Cellulitis (Infections and infestations) | 2 (3)
Infections and infestations - Other, Left foot soft tissue infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Perianal infection (Infections and infestations) | 1 (2)
Infections and infestations - Other, left leg infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, possible URI (Infections and infestations) | 1 (1)
Infections and infestations - Other, right leg cellulitis (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Irritability (General disorders) | 5 (6)
Libido decreased (Psychiatric disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 4 (7)
Localized edema (General disorders) | 1 (3)
Lung infection (Infections and infestations) | 3 (4)
Lymphocyte count decreased (Investigations) | 15 (64)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Muscle Spasm Legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, muscle spasm (legs) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 11 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Multicentric Castleman's disease
Nervous system disorders - Other, Neuropathy hands (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Neuropathy toes (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Spinal stenosis (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, intermittent dragging of R foot (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 27 (165)
Night sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain (General disorders) | 13 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (13)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9)
Pharyngitis (Infections and infestations) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 18 (53)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (53)
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, a URI rhinorrhea x3 days (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Upper respiratory infection (URI)
Respiratory, thoracic and mediastinal disorders - Other, a URI w/ congestion and rhinorrhea x3 days (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 4 (9)
Shivering (General disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Right leg cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, hand foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, warts on the left 2nd toe (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 6 (8)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stomal ulcer (Injury, poisoning and procedural complications) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Upper respiratory infection (Infections and infestations) | 8 (9)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight gain (Investigations) | 6 (6)
Weight loss (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 22 (100)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT01495598/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT01495598/ICF_001.pdf